CLINICAL TRIAL: NCT04331158
Title: The Effects of Dry Cupping on Pain, Function and Quality of Life of Women With Knee Osteoarthritis: Protocol for a Placebo-controlled Randomized Trial
Brief Title: Dry Cupping Therapy in Knee Osteoarthritis
Acronym: VentosaOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, PT, PhD., Adjunct Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFRNventosaOA
Record Dates: First submitted 2020-03-29; First posted 2020-04-02 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Osteo Arthritis Knee; Pain, Chronic; Pain
Keywords: Chronic pain; Traditional Chinese Medicine; Complementary Therapie
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: dry cupping group and dry cupping sham group
Who Masked: Participant, Outcomes Assessor
Masking Description: To avoid any type of selection bias, the confidential allocation method will be through opaque envelopes, sealed and numbered consecutively. The randomization process will be carried out by an independent researcher who will not be involved in other study procedures. The group in which the participant will be allocated will be revealed to the researcher responsible for the consultations prior to the first intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry cupping group (Experimental): The dry cupping will be applied with a force of two suctions generating a negative pressure on the skin during the time of 15 minutes.
  Interventions: Other: Dry cupping therapy
- Dry cupping sham group (Placebo Comparator): The dry cupping sham group will receive the same procedures as the dry cup group, with the difference that the negative pressure imposed after application will be released in a few seconds.
  Interventions: Other: Dry cupping therapy

INTERVENTIONS:
Other: Dry cupping therapy — Dry cupping therapy application on the patient's skin

SUMMARY:
Introduction: Knee osteoarthritis (KOA) is the biggest cause of pain and disability worldwide. As a non-pharmacological approach, ventosatherapia has been used to control pain, improve function and quality of life. However, there is a lack of high-quality scientific evidence regarding its effects on this condition. Objective: To evaluate the effects of dry cupping on pain, function and quality of life in women with KOA. Methods: This is a randomized, blinded placebo-controlled protocol. 62 women diagnosed with KOA will be recruited, based on the clinical criteria of the American College of Rheumatology, who will be randomly divided into two groups (31 per group): dry cupping and dry cupping sham.

DETAILED DESCRIPTION:
The intervention will be carried out for 15 minutes, twice a week, for 6 consecutive weeks, totaling 12 sessions. Both groups will be evaluated in 4 moments: before the intervention (T0), after 3 weeks of interventions (T3), at the end of the protocol (T6) and 4 weeks after the end of the interventions (follow-up - T10). The analyzed outcomes will be: Primary - pain (numerical pain scale); Secondary - Physical function (WOMAC; tests of going up / down stairs, brisk walking in 40 m and sitting / rising from a chair in 30 s), quality of life (SF-36) and global perception of the effect

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with KOA based on ACR clinical criteria;
* Knee pain intensity between 3 and 8, according to the Numerical Pain Scale (END);
* BMI less than 35 kg / m2.

Exclusion Criteria:

* Having undergone physical therapy treatment for the knee in the 3 months prior to the project;
* Be engaged in> 45 minutes / week in accumulated physical activity of at least moderate intensity;
* To have been submitted to the application and / or intervention with the wind therapy previously.
* Have used corticosteroid infiltration in the knee in the last 6 months;
* Present any medical restrictions that make it impossible for them to participate in the proposed assessments and interventions (cardiorespiratory, neurological and / or musculoskeletal changes);
* Presenting a diagnosis of fibromyalgia, rheumatoid arthritis or some systemic inflammatory arthritis;
* Presenting a ligament or meniscal injury diagnosed clinically or with a positive result in the Apley tests or anterior / posterior drawer;
* Have had previous surgery on the ankle, knee or hip;
* Present a clinical diagnosis of some dementia or inability to answer the questionnaires related to the study;
* Present any contraindications for the use of ventosatherapia (skin lesion in the region where it will be applied, cancer, kidney failure, liver and heart failure, pacemaker, pregnancy);
* Having uncontrolled diabetes and hypertension;
* Have a trip scheduled for the two months following inclusion in the survey.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Most prevalent disease in elderly women
Enrollment: 62 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Change from Numerical Rating Scale (NRS) | baseline, 3 ,6 and 10 weeks after.
  Subjective measure in which individuals rate their pain on an eleven-point numerical scale. Such scale will be positioned in front of the participant and will vary from 0 to 10 points, with 0 being the complete absence of pain and 10 being the worst pain imaginable by the individual

SECONDARY OUTCOMES:
Change from Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 3 ,6 and 10 weeks after.
  Questionnaire translated and validated for the Portuguese language, specific for the evaluation of patients with KOA, contains 24 questions divided into three categories that assess pain, stiffness and self-reported physical function.38 The items are evaluated by a Likert scale and each question receives a score that varies from 0 to 96 points, according to the patient's response (none = 0; low = 1; moderate = 2; severe = 3; very severe = 4). The higher the score obtained, the worse the severity of pain, stiffness or physical function
Change from 30-second Chair Stand Test | baseline, 6 and 10 weeks after.
  The sit and stand test will be performed in a chair without armrests, with a height of 43 cm, with non-slip rubber under its four supports. The back of the chair will be supported by a wall to prevent oscillations during the movements of sitting and standing. The participant will sit in the middle of the chair, with an erect back, feet apart and aligned with the joints of the respective shoulders and supported on a flat and stable floor. The test will consist of getting up from the chair as many times as possible, for 30 seconds. In this way, it will be possible to assess different levels of skill, with scores ranging from 0, for those who cannot complete a single repetition, to values greater than 20 repetitions, for the most able and well-prepared individuals
Change from 8-step Stair Climb Test | baseline, 6 and 10 weeks after.
  In the test of going up and down stairs, the participant will be positioned in front of the stairs and, at the signal, must go up the indicated steps (8 steps) and go down, in the shortest time possible. The height of each step will be 20 cm and it will be a staircase with a handrail, in a lighted environment, free of traffic and external distractions. A pre-test will be carried out to identify the need for security measures. The final score will be calculated based on the time the participant performed the procedure and compared with normative values available for the test.
Change from 40m Fast Paced Walk Test | baseline, 6 and 10 weeks after.
  The 40 meter fast walk test will be performed on 4 circuits of 10 meters (marked by ribbons and bounded by cones), in which the participant will be guided to walk the 10 meters, go around the cone and travel the next 10 meters again, successively, until the total distance of 40 meters is completed. The time will be timed only between the markings (start and end). The final score will be calculated based on the time the participant will perform the procedure and compared with normative values for healthy adults.
Change from Short-Form 36 quality of life | baseline, 6 and 10 weeks after.
  The instrument consists of 36 questions and assesses eight different domains that influence quality of life, considering the individual's perception of aspects of his health in the past weeks. Each item has a group of responses distributed on a graduated Likert scale, with the following dimensions: physical function, physical aspect, pain, general health, vitality, social function, emotional aspect and mental health. Your total score ranges from 0 to 100, where the higher the value, the better the quality of life.
Change from Global Perceived Effect | baseline, 3, 6 and 10 weeks after.
  Global perceived effect (GPE) is a 11-point Likert scale (ranging from -5 to +5) that compares the patients' current health status with that at the onset of symptoms. Positive scores are attributed to individuals who improved when compared with baseline and negative scores to those who worsened
Change from use of analgesics and anti-inflammatories | baseline, 3, 6 and 10 weeks after
  Number of use of analgesics and anti-inflammatories at the end of the study.
Change from expectation with treatment after the intervention protocol . | baseline and 10 weeks after
  A 5-point Likert scale was applied to assess patient expectation in terms of the intervention. The scale will be placed in front of the participant, who will be asked the following question: 'with dry cupping intervention do you think your situation will: (1) worsen considerably, (2) worsen a little, (3) neither improve nor worsen, (4) improve a little or (5) improve considerably

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo C de Souza, PT, PhD, Study Chair — Universidade Federal do Rio Grande do Norte
Locations (1):
- Marcelo Cardoso de Souza, Santa Cruz, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
there is not a plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Silva HJA, Saragiotto BT, Silva RS, Lins CAA, de Souza MC. Dry cupping in the treatment of individuals with non-specific chronic low back pain: a protocol for a placebo-controlled, randomised, double-blind study. BMJ Open. 2019 Dec 22;9(12):e032416. doi: 10.1136/bmjopen-2019-032416. PMID 31871257
- [Background] Peat G, Thomas E, Duncan R, Wood L, Hay E, Croft P. Clinical classification criteria for knee osteoarthritis: performance in the general population and primary care. Ann Rheum Dis. 2006 Oct;65(10):1363-7. doi: 10.1136/ard.2006.051482. Epub 2006 Apr 20. PMID 16627539
- [Derived] Cavalcanti RR, Almeida Silva HJ, Pontes-Silva A, Avila MA, de Souza CG, Sousa CO, Scattone Silva R, Barbosa GM, de Souza MC. Dry cupping therapy has no effect on pain, function, or quality of life in women with knee osteoarthritis: Randomized placebo-controlled trial. Braz J Phys Ther. 2026 Jan-Feb;30(1):101259. doi: 10.1016/j.bjpt.2025.101259. Epub 2025 Oct 2. PMID 41043303
- [Derived] Pontes NS, Barbosa GM, Almeida Silva HJ, Scattone Silva R, Souza CG, Lins CAA, de Souza MC. Effects of dry cupping on pain, function and quality of life in women with knee osteoarthritis: a protocol for a sham-controlled randomised trial. BMJ Open. 2020 Dec 24;10(12):e039857. doi: 10.1136/bmjopen-2020-039857. PMID 33361075